CLINICAL TRIAL: NCT04505722
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study to Assess the Efficacy and Safety of Ad26.COV2.S for the Prevention of SARS-CoV-2-mediated COVID-19 in Adults Aged 18 Years and Older
Brief Title: A Study of Ad26.COV2.S for the Prevention of SARS-CoV-2-Mediated COVID-19 in Adult Participants
Acronym: ENSEMBLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR108876; VAC31518COV3001 (Other: Janssen Vaccines & Prevention B.V.)
Expanded Access: NCT04817657 (No longer available)
Record Dates: First submitted 2020-07-31; First posted 2020-08-10 (Actual); Results first posted 2022-04-15 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Participants With or Without Stable Co-morbidities Associated With Progression to Severe COVID-19 at Different Stages of the Protocol
Keywords: Prevention; Vaccine
MeSH Terms: interventions — Ad26COVS1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ad26.COV2.S (Experimental): Participants will receive intramuscular (IM) injection of Ad26.COV2.S at a dose level of 5*10^10 virus particles (vp) as single dose vaccine on Day 1. At Year 1 (booster visit), participants who previously received any coronavirus disease-2019 (COVID-19) vaccination (as primary regimen or additional dose) will be offered a single booster dose of Ad26.COV2.S at the 5*10^10 vp dose level.
  Interventions: Biological: Ad26.COV2.S
- Placebo (Experimental): Participants will receive IM injection of placebo on Day 1. At Month 6/unblinding visit, post Emergency Use Authorization (EUA), conditional licensure, or approval for the single dose regimen, participants initially receiving placebo will be offered to receive a single dose of Ad26.COV2.S vaccine IM at a dose level of 5*10^10 vp. At Year 1 (booster visit), participants who previously received any COVID-19 vaccination (as primary regimen or additional dose) will be offered a single booster dose of Ad26.COV2.S at the 5*10^10 vp dose level.
  Interventions: Biological: Ad26.COV2.S; Other: Placebo

INTERVENTIONS:
Biological: Ad26.COV2.S — Ad26.COV2.S will be administered at a single dose of 5*10^10 virus particles (vp) on Day 1 (or Month 6 for placebo recipients) and as a single booster dose at Year 1.
  Other Names: JNJ-78436735; Ad26COVS1
Other: Placebo — Participants will receive Placebo.
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy of Ad26.COV2.S in the prevention of molecularly confirmed moderate to severe/critical COVID-19, as compared to placebo, in adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Contraceptive (birth control) use should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies
* All participants of childbearing potential must: have a negative highly sensitive urine pregnancy test at screening; and have a negative highly sensitive urine pregnancy test immediately prior to each study vaccine administration
* Participant agrees to not donate bone marrow, blood, and blood products from the first study vaccine administration until 3 months after receiving the last dose of study vaccine
* Must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study
* Must be able to read, understand, and complete questionnaires in the electronic clinical outcome assessment (eCOA) (that is, the coronavirus disease-2019 [COVID 19] signs and symptoms surveillance question, the e-Diary, and the electronic patient-reported outcomes (ePROs). Note: Participants with visual impairment are eligible for study participation and may have caregiver assistance in completing the electronic clinical outcome assessment (eCOA) questionnaires

Exclusion Criteria:

* Participant has a clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature greater than or equal to (>=) 38.0 degree Celsius (100.4-degree Fahrenheit) within 24 hours prior to the planned first dose of study vaccine; randomization at a later date is permitted at the discretion of the investigator and after consultation with the sponsor
* Participant received or plans to receive: (a) licensed live attenuated vaccines - within 28 days before or after planned administration of study vaccine ; and (b) other licensed (not live) vaccines - within 14 days before or after planned administration of study vaccine
* Participant previously received a coronavirus vaccine
* Participant received an investigational drug (including investigational drugs for prophylaxis of COVID-19) within 30 days or used an invasive investigational medical device within 30 days or received investigational immunoglobulin (Ig) or monoclonal antibodies within 3 months, or received convalescent serum for COVID-19 treatment within 4 months or received an investigational vaccine (including investigational Adenoviral-vectored vaccines) within 6 months before the planned administration of the first dose of study vaccine or is currently enrolled or plans to participate in another investigational study during the course of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44325 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (224):
- United States (117):
  - Synexus Clinical Research US Inc, Birmingham, Alabama
  - University of Alabama Birmingham, Birmingham, Alabama
  - Alabama Vaccine Research Clinic at UAB, Birmingham, Alabama
  - Optimal Research, Huntsville, Alabama
  - Synexus Clinical Research US Inc, Glendale, Arizona
  - VA Medical Center, Phoenix, Arizona
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Quality of Life Medical & Research Center, LLC, Tucson, Arizona
  - Synexus Clinical Research US Inc, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Ark Clinical Research, Long Beach, California
  - Anthony Mills Medical, Inc, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - UCSD Antiviral Research Center AVRC, San Diego, California
  - Wr McCr Llc, San Diego, California
  - VA Medical Center, San Francisco, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Regional VA Medical Center, Denver, Colorado
  - Avail Clinical Research, LLC, DeLand, Florida
  - North Florida South Georgia Veteran Health System, Gainesville, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Research Centers of America, LLC, Hollywood, Florida
  - Suncoast Research Group, Miami, Florida
  - University of Miami - Miller School of Medicine, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Advent Health Orlando, Orlando, Florida
  - Synexus Clinical Research US Inc, Orlando, Florida
  - Synexus Clinical Research US Inc, Pinellas Park, Florida
  - James A Haley VA Hospital GNS, Tampa, Florida
  - Synexus Clinical Research US Inc, The Villages, Florida
  - Emory University of Medicine, Atlanta, Georgia
  - The Hope Clinic at Emory University, Decatur, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northwestern University, Chicago, Illinois
  - Jesse Brown VAMC Department of Surgery, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of IL Chicago, Chicago, Illinois
  - The University Of Chicago Medicine, Chicago, Illinois
  - Optimal Research, Peoria, Illinois
  - Buynak Clinical Research, Valparaiso, Indiana
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Benchmark Research, Metairie, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - New Orleans Adolescent Trials Unit CRS, New Orleans, Louisiana
  - Southeast Louisiana Veterans Health Care Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Baltimore VA Medical Center, Baltimore, Maryland
  - Optimal Research, Rockville, Maryland
  - Meridian Clinical Research, LLC, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Brigham and Women's Hospital, Inc., Boston, Massachusetts
  - University of Michigan Neuorsurgery A. Alfred Taubman Health Care Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Cherry Street Services, Inc., Grand Rapids, Michigan
  - Abbott Northwestern Hospital Clinic, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - MediSync Clinical Research, Petal, Mississippi
  - The Center For Pharmaceutical Research, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Synexus Clinical Research US Inc, St Louis, Missouri
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Clinical Research Consortium, an AMR company, Las Vegas, Nevada
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Saint Michaels Medical Center, Newark, New Jersey
  - Raymond G. Murphy VA Medical Center, Albuquerque, New Mexico
  - Meridian Clinical Research, LLC, Endwell, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Harlem Hospital Center, New York, New York
  - New York Blood Center, New York, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Bronx Veterans Affairs Medical Center, The Bronx, New York
  - Tryon Medical Group, Charlotte, North Carolina
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Durham VAMC, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Synexus Clinical Research US Inc, Akron, Ohio
  - CTI Clinical Trial and Consulting Services, Cincinnati, Ohio
  - Synexus Clinical Research US Inc, Cincinnati, Ohio
  - Velocity Clinical Research, Cincinnati, Ohio
  - Rapid Medical Research, Cleveland, Ohio
  - Synexus Clinical Research US Inc, Columbus, Ohio
  - Corvallis Clinic PC, Corvallis, Oregon
  - Clinical Research Institute of Southern Oregon, P.C., Medford, Oregon
  - Oregon Health And Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Synexus Clinical Research US Inc, Anderson, South Carolina
  - VA Medical Center, Columbia, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - PMG Research of Charleston, LLC, Mt. Pleasant, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Benchmark Research, Austin, Texas
  - Optimal Research, LLC, Austin, Texas
  - AIDS Arms Incorporated Trinity Health and Wellness Center, Dallas, Texas
  - Synexus Clinical Research US Inc, Dallas, Texas
  - Baylor Scott and White Research Institute, Dallas, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Texas Center for Drug Development Inc, Houston, Texas
  - Gordon Crofoot, MD, Houston, Texas
  - Clinical Trials of Texas Inc, San Antonio, Texas
  - Synexus Clinical Research US Inc, San Antonio, Texas
  - Synexus Clinical Research US Inc, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington
- Argentina (12):
  - Clínica y Maternidad Suizo Argentina, Buenos Aires
  - CIPREC, Buenos Aires
  - Helios Salud Sa, Buenos Aires
  - CEMEDIC, Buenos Aires
  - Centro Medico Viamonte SRL, Ciudad Autonoma Buenos Aires
  - Clinical Trials Division-Stamboulian Servicios de Salud, Ciudad Autonoma Buenos Aires
  - Fundacion Huesped, Ciudad Autonoma de Buenos Aire
  - CEMIC Saavedra, Ciudad de Buenos Aires
  - Hospital J. M. Ramos Mejía, Ciudad de Buenos Aires
  - Instituto Medico Platense, La Plata
  - Hospital Italiano de La Plata, La Plata
  - DIM Clinica Privada, Ramos Mejía
- Brazil (27):
  - Faculdade de Medicina Barretos FACISB, Barretos
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - L2IP Instituto de Pesquisas Clinicas, Brasília
  - Sociedade Campineira de Educacao e Instrucao Hospital e Maternidade Celso Pierro, Campinas
  - Fundacao Universidade Federal de Mato Grosso do Sul, Campo Grande
  - Sociedade Literaria e Caritativa Santo Agostinho Hospital Sao Jose, Criciúma
  - Oncovida - Centro de Onco-Hematologia de Mato Grosso, Cuiabá
  - Hospital Nossa Senhora Das Gracas, Curitiba
  - Centro de Estudos e Pesquisas em Moléstias Infecciosas, Natal
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Hospital Nossa Senhora da Conceicao S A, Porto Alegre
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Ministerio da Saude - Hospital dos Servidores do Estado - RJ, Rio de Janeiro
  - Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
  - Fundacao Oswaldo Cruz, Rio de Janeiro
  - Municipio de Nova Iguacu - Hospital Geral de Nova Iguacu, Rio de Janeiro
  - Fundacao Bahiana De Infectologia, Salvador
  - Universidade Municipal de Sao Caetano do Sul, São Caetano do Sul
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - CPQuali Pesquisa Clinica LTDA ME, São Paulo
  - Instituto de infectologia Emilio Ribas, São Paulo
  - Sociedade Beneficente de Senhoras - Hospital Sírio Libanês, São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
  - Centro de Referencia E Treinamento Dst/Aids, São Paulo
  - CEPIC Centro Paulista de Investigacao Clinica e Servicos Medicos, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Chile (6):
  - Centro de Estudios Clínicos e Investigación Médica (CeCim), Santiago
  - Facultad de Medicina Universidad de Chile, Santiago
  - Hospital Padre Hurtado, Santiago
  - Centro de Investigacion del Maule, Talca
  - Hospital Dr Hernan Henriquez Aravena, Temuco
  - Centro de Estudios Clinicos V Region Ltda, Viña del Mar
- Colombia (13):
  - Clinica de la Costa, Barranquilla
  - Centro de Reumatologia y Ortopedia, Barranquilla
  - Hospital Universidad del Norte, Barranquilla
  - Centro de Atencion e Investigacion Medica S.A. - CAIMED, Bogotá
  - Medplus Medicina Prepagada S.A., Bogotá
  - Solano y Terront Servicios Médicos Ltda., Bogotá
  - Centro de Investigaciones Clinicas S A S, Cali
  - Fundación Valle del Lili, Cali
  - Fundación Cardiovascular de Colombia - Instituto del Corazón Floridablanca, Floridablanca
  - Fundacion Oftalmologica de Santander - FOSCAL, Floridablanca
  - Programa de Estudio y Control de Enfermedades Tropicales, Medellín
  - Hospital Pablo Tobon Uribe, Medellín
  - Fundacion Centro de Investigacion Clinica CIC, Medellín
- Mexico (9):
  - Instituto Nacional de Salud Publica, Cuernavaca
  - Hospital Civil Fray Antonio Alcalde, Guadalajara
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Unidad de Atención Medica e Investigacion en Salud (UNAMIS), Mérida
  - Centro Medico Nacional Siglo XXI IMSS, México
  - CAIMED Investigacion en salud S.A de C.V., México
  - Instituto Nacional de Enfermedades Respiratorias, México
  - Hospital Universitario de Nuevo Leon 'Dr Jose Eleuterio Gonzalez', Monterrey
  - Infectolab, Tijuana
- Peru (10):
  - Centro de Invetigaciones Medicas, Callao
  - Hospital Nacional Daniel Alcides Carrion, Callao
  - Centro de Investigaciones Tecnologicas, Biomedica y medio ambientales (CITBM), Callao
  - Asociacion Civil Selva Amazonica (ACSA), Iquitos
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
  - Hospital Nacional Arzobispo Loayza, Lima
  - Asociacion Civil Via Libre, Lima
  - Instituto de Investigacion Nutricional, Lima
  - Asociacion Civil Impacta Salud y Educacion- San Miguel CRS, Lima
  - Asociacion Civil Impacta Salud y Educacion - Barranco, Lima - Barranco
- South Africa (30):
  - Josha Research, Bloemfontein
  - Synexus Helderberg Clinical Research Centre, Cape Town
  - Family Clinical Research Unit FAM-CRU, Cape Town
  - TASK Central, Cape Town
  - Desmond Tutu HIV Foundation, Cape Town
  - University of Cape Town IDM/CIDRI Research Site, Cape Town
  - Desmond Tutu Hiv Foundation - University Of Cape Town, Cape Town
  - Masiphumelele Research Centre, Cape Town
  - Ndlovu Elandsdoorn Site, Dennilton
  - SA Medical Research Council, Durban
  - CRISMO Bertha Gxowa Research Centre, Johannesburg
  - Shandukani Research Centre, Johannesburg
  - The Aurum Institute Klerksdorp Clinical Research Centre, Klerksdorp
  - Qhakaza Mbokodo Research Centre, KwaZulu-Natal
  - South African Medical Research Council Chatsworth Clinical Research Site, KwaZulu-Natal
  - Centre for the AIDS Programme of Research in South Africa, KwaZulu-Natal
  - Stanza Clinical Research Centre : Mamelodi, Mamelodi East
  - Mzansi Ethical Research Centre, Middelburg
  - Nelson Mandela Academic Clinical Research Unit 'NeMACRU', Mthatha
  - PHOENIX PHARMA (Pty) Ltd, Port Elizabeth
  - MeCRU Clinical Research Unit, Pretoria
  - Synexus Watermeyer, Pretoria
  - The Aurum Institute Rustenburg Clinical Research Site, Rustenburg
  - Setshaba Research Centre, Soshanguve
  - Perinatal HIV Research Unit (PHRU), Kliptown, Soweto
  - Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital, Soweto
  - The Aurum Institute: Tembisa - Clinic 4, Tembisa
  - CAPRISA Vulindlela Clinic, Vulindlela
  - University of Witwatersrand - Helen Joseph Hospital - Themba Lethu Hiv Research Centre, Westdene Johannesburg Gauteng
  - SATVI, Brewelskloof Hospital, Worcester

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Carpp LN, Hyrien O, Fong Y, Benkeser D, Roels S, Stieh DJ, Van Dromme I, Van Roey GA, Kenny A, Huang Y, Carone M, McDermott AB, Houchens CR, Martins K, Jayashankar L, Castellino F, Amoa-Awua O, Basappa M, Flach B, Lin BC, Moore C, Naisan M, Naqvi M, Narpala S, O'Connell S, Mueller A, Serebryannyy L, Castro M, Wang J, Petropoulos CJ, Luedtke A, Lu Y, Yu C, Juraska M, Hejazi NS, Wolfe DN, Sadoff J, Gray GE, Grinsztejn B, Goepfert PA, Bekker LG, Gaur AH, Veloso VG, Randhawa AK, Andrasik MP, Hendriks J, Truyers C, Vandebosch A, Struyf F, Schuitemaker H, Douoguih M, Kublin JG, Corey L, Neuzil KM, Follmann D, Koup RA, Donis RO, Gilbert PB; Immune Assays Team; Coronavirus Vaccine Prevention Network (CoVPN)/ENSEMBLE Team; United States Government (USG)/CoVPN Biostatistics Team. Neutralizing antibody correlate of protection against severe-critical COVID-19 in the ENSEMBLE single-dose Ad26.COV2.S vaccine efficacy trial. Nat Commun. 2024 Nov 12;15(1):9785. doi: 10.1038/s41467-024-53727-y. PMID 39532861
- [Derived] Janes H, Fisher LH, Kee JJ, Parameswaran L, Goepfert PA, Falsey AR, Ludwig J, Magaret CA, Gilbert PB, Kublin JG, Rouphael N, Sobieszczyk ME, El Sahly HM, Baden LR, Grinsztejn B, Walsh SR, Gray GE, Kotloff KL, Gay CL, Greninger AL, Tapia MD, Hammershaimb EA, Priddy FH, Green JA, Struyf F, Dunkle L, Neuzil KM, Corey L, Huang Y. Association Between SARS-CoV-2 Viral Load and COVID-19 Vaccination in 4 Phase 3 Trials. J Infect Dis. 2024 Dec 16;230(6):1384-1389. doi: 10.1093/infdis/jiae400. PMID 39225478
- [Derived] Turley CB, Tables L, Fuller T, Sanders LJ, Scott H, Moodley A, Woodward Davis A, Leav B, Miller J, Schoemaker K, Vandebosch A, Sadoff J, Woo W, Cho I, Dunkle LM, Li S, van der Laan L, Gilbert PB, Follmann D, Jaynes H, Kublin JG, Baden LR, Goepfert P, Kotloff K, Gay CL, Falsey AR, El Sahly HM, Sobieszczyk ME, Huang Y, Neuzil KM, Corey L, Grinsztejn B, Gray G, Rouphael N, Luedtke A; COVID-19 Prevention Network CoVPN. Modifiers of COVID-19 vaccine efficacy: Results from four COVID-19 prevention network efficacy trials. Vaccine. 2023 Jul 25;41(33):4899-4906. doi: 10.1016/j.vaccine.2023.06.066. Epub 2023 Jun 23. PMID 37385888
- [Derived] Fong Y, McDermott AB, Benkeser D, Roels S, Stieh DJ, Vandebosch A, Le Gars M, Van Roey GA, Houchens CR, Martins K, Jayashankar L, Castellino F, Amoa-Awua O, Basappa M, Flach B, Lin BC, Moore C, Naisan M, Naqvi M, Narpala S, O'Connell S, Mueller A, Serebryannyy L, Castro M, Wang J, Petropoulos CJ, Luedtke A, Hyrien O, Lu Y, Yu C, Borate B, van der Laan LWP, Hejazi NS, Kenny A, Carone M, Wolfe DN, Sadoff J, Gray GE, Grinsztejn B, Goepfert PA, Little SJ, Paiva de Sousa L, Maboa R, Randhawa AK, Andrasik MP, Hendriks J, Truyers C, Struyf F, Schuitemaker H, Douoguih M, Kublin JG, Corey L, Neuzil KM, Carpp LN, Follmann D, Gilbert PB, Koup RA, Donis RO; Immune Assays Team; Coronavirus Vaccine Prevention Network (CoVPN)/ENSEMBLE Team; and the United States Government (USG)/CoVPN Biostatistics Team. Immune correlates analysis of the ENSEMBLE single Ad26.COV2.S dose vaccine efficacy clinical trial. Nat Microbiol. 2022 Dec;7(12):1996-2010. doi: 10.1038/s41564-022-01262-1. Epub 2022 Nov 10. PMID 36357712
- [Derived] Sadoff J, Gray G, Vandebosch A, Cardenas V, Shukarev G, Grinsztejn B, Goepfert PA, Truyers C, Van Dromme I, Spiessens B, Vingerhoets J, Custers J, Scheper G, Robb ML, Treanor J, Ryser MF, Barouch DH, Swann E, Marovich MA, Neuzil KM, Corey L, Stoddard J, Hardt K, Ruiz-Guinazu J, Le Gars M, Schuitemaker H, Van Hoof J, Struyf F, Douoguih M; ENSEMBLE Study Group. Final Analysis of Efficacy and Safety of Single-Dose Ad26.COV2.S. N Engl J Med. 2022 Mar 3;386(9):847-860. doi: 10.1056/NEJMoa2117608. Epub 2022 Feb 9. PMID 35139271
- [Derived] Sadoff J, Struyf F, Douoguih M. A plain language summary of how well the single-dose Janssen vaccine works and how safe it is. Future Virol. 2021 Nov;16(11):725-739. doi: 10.2217/fvl-2021-0199. Epub 2021 Nov 1. PMID 34824596
- [Derived] Sadoff J, Gray G, Vandebosch A, Cardenas V, Shukarev G, Grinsztejn B, Goepfert PA, Truyers C, Fennema H, Spiessens B, Offergeld K, Scheper G, Taylor KL, Robb ML, Treanor J, Barouch DH, Stoddard J, Ryser MF, Marovich MA, Neuzil KM, Corey L, Cauwenberghs N, Tanner T, Hardt K, Ruiz-Guinazu J, Le Gars M, Schuitemaker H, Van Hoof J, Struyf F, Douoguih M; ENSEMBLE Study Group. Safety and Efficacy of Single-Dose Ad26.COV2.S Vaccine against Covid-19. N Engl J Med. 2021 Jun 10;384(23):2187-2201. doi: 10.1056/NEJMoa2101544. Epub 2021 Apr 21. PMID 33882225
- [Derived] Williams TC, Burgers WA. SARS-CoV-2 evolution and vaccines: cause for concern? Lancet Respir Med. 2021 Apr;9(4):333-335. doi: 10.1016/S2213-2600(21)00075-8. Epub 2021 Jan 29. No abstract available. PMID 33524316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 44325 participants were randomized, of which 1 participant was randomized in error due to lack of a signed informed consent form. This participant has not been included in the analysis.
Pre-assignment Details: Due to change in the planned analysis, combined data of "double blind (DB)" and "open label (OL)" phase was collected and analyzed after completion of the double-blind phase. Results of safety outcome measures (OMs) were also collected and analyzed for combined DB and OL phase. Hence, safety data is reported only in adverse event section and not repeated in the OMs section. In all-cause mortality section out of 324 deaths, 1 death was not related to Adverse event.
Groups:
- Double-blind Phase: Ad26.COV2.S 5*10^10 vp: Participants received intramuscular (IM) injection of Ad26.COV2.S at a dose level of 5*10^10 virus particles (vp) as single dose vaccine on Day 1.
- Double-blind Phase: Placebo: Participants received IM injection of placebo matching to Ad26.COV2.S on Day 1.
- Combined Double-blind and Open-label Phase: All Participants: Participants received a single dose of Ad26.COV2.S 5*10^10 vp vaccine or placebo as IM injection on Day 1. At Month 6/unblinding visit, post emergency use authorization (EUA), conditional licensure, or approval for the single dose regimen, participants initially receiving placebo were offered a single dose of Ad26.COV2.S vaccine IM at a dose level of 5*10^10 vp. As of implementation of protocol amendment 3, participants were allowed to have an outside COVID-19 vaccine. As of implementation of protocol amendment 6, at Year 1 (open label booster vaccination phase), participants who previously received any COVID-19 vaccine (as primary regimen or additional dose) with the Ad26.COV2.S vaccine, and/or an mRNA vaccine or another COVID-19 vaccine authorized for primary vaccination were offered a single booster dose of Ad26.COV2.S at the 5*10^10 vp dose level.
Period: DB Phase (Day 1 up to 6 Months)
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo | Combined Double-blind and Open-label Phase: All Participants
Started | 22174 | 22150 | 0
Vaccinated | 21898 | 21890 | 0
Completed | 21138 | 20662 | 0
Not Completed | 1036 | 1488 | 0
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Death | 34 | 63 | 0
Not completed — Lost to Follow-up | 271 | 333 | 0
Not completed — Physician Decision | 17 | 17 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 376 | 714 | 0
Not completed — Other | 61 | 98 | 0
Not completed — Randomized not vaccinated | 276 | 260 | 0
Period: DB + OL Phase (2 Years 6.5 Months)
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo | Combined Double-blind and Open-label Phase: All Participants
Started | 0 | 0 | 43788 (Only vaccinated participants of combined double blind and open label phase are included in the analysis.)
Completed | 0 | 0 | 31593
Not Completed | 0 | 0 | 12195
Not completed — Adverse Event | 0 | 0 | 6
Not completed — Death | 0 | 0 | 324
Not completed — Lost to Follow-up | 0 | 0 | 4978
Not completed — Physician Decision | 0 | 0 | 342
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 4332
Not completed — Other | 0 | 0 | 2211

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants with a documented double-blind study vaccine administration, regardless of the occurrence of protocol deviations and serostatus at enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo | Total
Number analyzed (Participants) | 21898 | 21890 | 43788
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (15.08) | 50.7 (15.04) | 50.7 (15.06)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 9828 | 9907 | 19735
  Male | 12067 | 11979 | 24046
  Undifferentiated | 2 | 4 | 6
  Unknown | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9875 | 9964 | 19839
  Not Hispanic or Latino | 11476 | 11367 | 22843
  Unknown or Not Reported | 547 | 559 | 1106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2083 | 2060 | 4143
  Asian | 743 | 686 | 1429
  Native Hawaiian or Other Pacific Islander | 56 | 47 | 103
  Black or African American | 4253 | 4262 | 8515
  White | 12858 | 12843 | 25701
  More than one race | 1207 | 1248 | 2455
  Unknown or Not Reported | 698 | 744 | 1442
Region of Enrollment [Number; unit: participants]
  ARGENTINA | 1498 | 1498 | 2996
  BRAZIL | 3644 | 3635 | 7279
  CHILE | 563 | 570 | 1133
  COLOMBIA | 2125 | 2123 | 4248
  MEXICO | 238 | 241 | 479
  PERU | 886 | 885 | 1771
  SOUTH AFRICA | 3287 | 3289 | 6576
  UNITED STATES | 9657 | 9649 | 19306

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of Molecularly Confirmed Moderate to Severe/Critical Coronavirus Disease (COVID-19) With Seronegative Status With Onset at Least 14 Days After Double-blind Vaccination on Day 1 (Day 15): Double-blind Phase
Description: Molecularly confirmed moderate to severe/critical COVID-19 was defined as a severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) positive reverse transcription/polymerase chain reaction (RT-PCR) or molecular test result from any available respiratory tract sample (example, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample. Moderate included one sign or symptom such as respiratory rate >= 20 breaths per minute and symptoms such as shortness of breath or two signs or symptoms such as heart rate >= 90 beats per minute (beats/minute) and symptoms such as cough from a list of signs and symptoms and severe/critical included one of the following signs and symptoms: respiratory rate >=30 breaths/minute, heart rate >=125 beats/minute, oxygen saturation (SpO2) <= 93% on room air at sea level respiratory failure, evidence of shock, significant acute renal, hepatic, or neurologic dysfunction, admission to the ICU, death defined as per FDA guidance.
Time Frame: From 14 days after double-blind vaccination on Day 1 (Day 15) up to Month 6
Population: Per-protocol Efficacy (PP) set: participants of the FAS (all randomized participants with double-blind study vaccine administration, regardless of protocol deviations and serostatus at enrollment) who received double-blind study vaccine and who were seronegative at the time of vaccination and who had no other major protocol deviations to possibly impact the efficacy of the vaccine. Participants who had a positive PCR test between Day 1 and Day 14 in PP set were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19400 | 19398
Participants
  Age: 18-59 years: number analyzed (Participants) | 12665 | 12674
  Age: 18-59 years | 381 | 847
  Age: Greater than or equal to (>=) 60 years: number analyzed (Participants) | 6735 | 6724
  Age: Greater than or equal to (>=) 60 years | 103 | 220

2. Primary Outcome: Number of Participants With First Occurrence of Molecularly Confirmed Moderate to Severe/Critical COVID-19 With Seronegative Status With Onset at Least 28 Days After Double-blind Vaccination on Day 1 (Day 29): Double-blind Phase
Description: Molecularly confirmed moderate to severe/critical COVID-19 was defined as a SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (example, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample. Moderate included one sign or symptom such as respiratory rate >=20 breaths per minute and symptoms such as shortness of breath or two signs or symptoms such as heart rate >= 90 beats/minute and symptoms such as cough from a list of signs and symptoms and severe/critical included one of the following signs and symptoms: respiratory rate >=30 breaths/minute, heart rate >=125 beats/minute, SpO2 less than or equal to (<=) 93 percent (%) on room air at sea level respiratory failure, evidence of shock, significant acute renal, hepatic, or neurologic dysfunction, admission to the Intensive Care Unit (ICU), death defined as per Food and Drug Administration (FDA) guidance.
Time Frame: From 28 days after double-blind vaccination on Day 1 (Day 29) up to Month 6
Population: PP set included participants of the Full Analysis Set (FAS) who received double-blind study vaccine and who were seronegative at the time of double-blind vaccination and who had no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine. Participants who had a positive PCR test between Day 1 and Day 28 in PP set were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19113 | 18924
Participants
  Age: 18-59 years: number analyzed (Participants) | 12489 | 12350
  Age: 18-59 years | 340 | 716
  Age: >=60 years: number analyzed (Participants) | 6624 | 6574
  Age: >=60 years | 93 | 167
  All participants | 433 | 883

3. Primary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) Up to 7 Days After Booster Vaccination (Open-label Booster Vaccination Phase)
Description: Participants who received the booster dose were asked to note in the e-Diary occurrences of injection site pain/tenderness, erythema, and swelling at the study vaccine injection site daily for 7 days post-booster vaccination (day of vaccination and the subsequent 7 days).
Time Frame: Up to Day 372 (7 Days after booster vaccination on Day 365 [Year 1])
Population: Full analysis booster set included all randomized participants with a documented study vaccine administration, regardless of the occurrence of protocol deviations and serostatus at enrollment, who received the Ad26.COV2.S booster vaccination at the booster visit.
Measure: Count of Participants; unit: Participants
Groups:
- OL Phase: Ad26.COV2.S 5*10^10 vp + Ad26.COV2.S 5*10^10 vp Booster: Participants received a single dose of Ad26.COV2.S 5*10^10 vp vaccine or placebo as IM injection on Day 1. At Month 6/unblinding visit, participants initially receiving placebo were offered a single dose of Ad26.COV2.S vaccine IM injection at a dose level of 5*10^10 vp. At Year 1 (booster visit), participants who previously received any COVID-19 vaccine (as primary regimen or additional dose) were offered a single booster dose of Ad26.COV2.S at the 5*10^10 vp dose level as booster vaccination.
- Open Label Phase: mRNA 2 Dose Schedule + Ad26.COV2.S 5*10^10 vp Booster: Participants who initially received a single dose of placebo vaccine matching to Ad26.COV2.S as IM injection on Day 1 in the double blind phase and received 2 doses of mRNA vaccination outside of the trial further received an Ad26.COV2.S booster dose at a dose level of 5*10^10 vp at 1 year after the initial vaccination, with a minimum of 3 months after the last outside vaccination.
- OL Phase: Non-mRNA Any Schedule +Ad26.COV2.S vp Booster OR mRNA Other Schedule +Ad26.COV2.S Booster: Participants who initially received a single dose of placebo vaccine matching to Ad26.COV2.S IM injection on Day 1 in double blind phase and received non-mRNA vaccination outside of the trial or only 1 dose of mRNA vaccination or more than 2 doses of mRNA vaccination further received an Ad26.COV2 booster dose at a dose level of 5*10^10 vp at 1 year after the initial vaccination, with a minimum of 3 months after the last outside vaccination.
Arm/Group | OL Phase: Ad26.COV2.S 5*10^10 vp + Ad26.COV2.S 5*10^10 vp Booster | Open Label Phase: mRNA 2 Dose Schedule + Ad26.COV2.S 5*10^10 vp Booster | OL Phase: Non-mRNA Any Schedule +Ad26.COV2.S vp Booster OR mRNA Other Schedule +Ad26.COV2.S Booster
Number analyzed (Participants) | 22213 | 613 | 943
Participants | 3758 | 135 | 204

4. Primary Outcome: Number of Participants With Solicited Systemic AEs Up to 7 Days After Booster Vaccination (Open-label Booster Vaccination Phase)
Description: Participants recorded the temperature in the e-Diary in the evening of the day of vaccination, and then daily for the next 7 days approximately at the same time each day. If more than 1 measurement was made on any given day, the highest temperature of that day was recorded in the e-Diary. Fever was defined as endogenous elevation of body temperature >= 38.0 degree Celsius or >=100.4-degree Fahrenheit, as recorded in at least 1 measurement. Participants also noted the signs and symptoms in the e-Diary on a daily basis for 7 days post-booster vaccination (day of vaccination and the subsequent 7 days), if feasible, for the following events: fatigue, headache, nausea, myalgia.
Time Frame: Up to Day 372 (7 Days after booster vaccination on Day 365 [Year 1])
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | OL Phase: Ad26.COV2.S 5*10^10 vp + Ad26.COV2.S 5*10^10 vp Booster | Open Label Phase: mRNA 2 Dose Schedule + Ad26.COV2.S 5*10^10 vp Booster | OL Phase: Non-mRNA Any Schedule +Ad26.COV2.S vp Booster OR mRNA Other Schedule +Ad26.COV2.S Booster
Number analyzed (Participants) | 22213 | 613 | 943
Participants | 3559 | 145 | 198

5. Primary Outcome: Number of Participants With Unsolicited AEs Up to 28 Days After Booster Vaccination (Open-label Booster Vaccination Phase)
Description: Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: Up to Day 393 (28 Days after booster vaccination on Day 365 [Year 1])
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | OL Phase: Ad26.COV2.S 5*10^10 vp + Ad26.COV2.S 5*10^10 vp Booster | Open Label Phase: mRNA 2 Dose Schedule + Ad26.COV2.S 5*10^10 vp Booster | OL Phase: Non-mRNA Any Schedule +Ad26.COV2.S vp Booster OR mRNA Other Schedule +Ad26.COV2.S Booster
Number analyzed (Participants) | 22213 | 613 | 943
Participants | 2133 | 58 | 95

6. Secondary Outcome: Number of Participants With First Occurrence of Molecularly Confirmed Severe/Critical COVID-19 With Seronegative Status With Onset at Least 14 Days After Double-blind Vaccination on Day 1 (Day 15): Double-blind Phase
Description: Molecularly confirmed severe/critical COVID-19 was defined as a SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (example, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample and one of the following signs and symptoms: respiratory rate >=30 breaths/minute, heart rate >=125 beats/minute,SpO2 <=93% on room air at sea level respiratory failure, evidence of shock, significant acute renal, hepatic, or neurologic dysfunction, admission to the ICU, death defined as per FDA guidance. Seronegative is defined as N-serology seronegative at the time of boosting or at the Year 1 visit if not boosted.
Time Frame: From 14 days after double-blind vaccination on Day 1 (Day 15) up to Month 6
Population: PP set included participants of the FAS who received double-blind study vaccine and who were seronegative at the time of double-blind vaccination and who had no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine. Participants who had a positive PCR test between Day 1 and Day 14 in PP set were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19400 | 19398
Participants | 56 | 205

7. Secondary Outcome: Number of Participants With First Occurrence of Molecularly Confirmed Severe/Critical COVID-19 With Seronegative Status With Onset at Least 28 Days After Double-blind Vaccination on Day 1 (Day 29): Double-blind Phase
Description: Severe/critical COVID-19 was defined as a SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (example, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample and one of the following signs and symptoms: respiratory rate >=30 breaths/minute, heart rate >=125 beats/minute,SpO2 <=93% on room air at sea level respiratory failure, evidence of shock, significant acute renal, hepatic, or neurologic dysfunction, admission to the ICU, death defined as per FDA guidance.
Time Frame: From 28 days after double-blind vaccination on Day 1 (Day 29) up to Month 6
Population: PP set included participants of the FAS who received double-blind study vaccine and who were seronegative at the time of double-blind vaccination and who had no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine. Participants who had a positive PCR test between Day 1 and Day 28 in PP set were excluded. Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19113 | 18924
Participants | 46 | 176

8. Secondary Outcome: Number of Participants With First Occurrence of Molecularly Confirmed Moderate to Severe/Critical COVID-19 Regardless of Their Serostatus (Double Blind Phase)
Description: Molecularly confirmed moderate to severe/critical COVID-19 was defined as a SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (example, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample. Moderate included one sign or symptom such as respiratory rate >= 20 breaths per minute and symptoms such as shortness of breath or two signs or symptoms such as heart rate >= 90 beats per minute (beats/minute) and symptoms such as cough from a list of signs and symptoms and severe/critical included one of the following signs and symptoms: respiratory rate >=30 breaths/minute, heart rate >=125 beats/minute,SpO2 <=93% on room air at sea level respiratory failure, evidence of shock, significant acute renal, hepatic, or neurologic dysfunction, admission to the ICU, death defined as per FDA guidance.
Time Frame: 1 day after double-blind vaccination on Day 1 (Day 2)
Population: FAS included all randomized participants with a documented double-blind study vaccine administration, regardless of the occurrence of protocol deviations and serostatus at enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 21898 | 21890
Participants | 575 | 1189

9. Secondary Outcome: Number of Participants With First Occurrence of Molecularly Confirmed Moderate to Severe/Critical COVID-19 Regardless of Their Serostatus (Double Blind Phase)
Description: as for outcome 8
Time Frame: 14 days after double-blind vaccination on Day 1 (Day 15)
Population: PP set included participants of the FAS who received double-blind study vaccine, regardless of their serostatus at the time of double-blind vaccination and who had no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine. This excludes participants who had a COVID-19 case with an onset before Day 15.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 21537 | 21467
Participants | 487 | 1079

10. Secondary Outcome: Number of Participants With First Occurrence of Molecularly Confirmed Moderate to Severe/Critical COVID-19 Regardless of Their Serostatus (Double Blind Phase)
Description: as for outcome 8
Time Frame: 28 days after double-blind vaccination on Day 1 (Day 29)
Population: PP set included participants of the FAS who received double-blind study vaccine, regardless of their serostatus at the time of double-blind vaccination and who had no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine. This excludes participants who had a COVID-19 case with an onset before Day 29.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 21244 | 20978
Participants | 436 | 895

11. Secondary Outcome: Number of Participants With First Occurrence of COVID-19 Requiring Medical Intervention (Double Blind Phase)
Description: Number of participants with first occurrence of COVID-19 requiring medical intervention (such as a composite endpoint of hospitalization, ICU admission, mechanical ventilation, and extracorporeal membrane oxygenation [ECMO], linked to objective measures such as decreased oxygenation, X-ray or computed tomography [CT] findings) or linked to any molecularly confirmed, COVID-19 at least 14 days post vaccination were reported.
Time Frame: 14 days after double-blind vaccination on Day 1 (Day 15)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19400 | 19398
Participants | 18 | 74

12. Secondary Outcome: Number of Participants With First Occurrence of COVID-19 Requiring Medical Intervention (Double Blind Phase)
Description: Number of participants with first occurrence of COVID-19 requiring medical intervention (such as a composite endpoint of hospitalization, ICU admission, mechanical ventilation, and ECMO, linked to objective measures such as decreased oxygenation, X-ray or CT findings) or linked to any molecularly confirmed, COVID-19 at least 28 days post vaccination were reported.
Time Frame: 28 Days after double-blind vaccination on Day 1 (Day 29)
Population: PP set included participants of the FAS who received double-blind study vaccine and who were seronegative at the time of double-blind vaccination and who had no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine. Participants who had a positive PCR test between Day 1 and Day 28 in PP set were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19113 | 18924
Participants | 16 | 64

13. Secondary Outcome: Area Under the Curve (AUC) of SARS-CoV-2 Viral Load as Assessed by Quantitative Reverse-Transcriptase Polymerase Chain Reaction (RT-PCR) in Participants With Molecularly Confirmed, Moderate to Severe/Critical COVID-19 (Double Blind Phase)
Description: AUC of SARS-CoV-2 Viral Load was assessed in confirmed COVID-19 cases using RT-PCR. Nasal swabs were used to detect and/or quantify SARS-CoV-2.
Time Frame: From Day 15 to end of the COVID-19 episode (Day 189)
Population: PP set included participants of the FAS who received double-blind study vaccine and who were seronegative at the time of double-blind vaccination and who had no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine. Participants who had a positive PCR test between Day 1 and Day 14 in PP set were excluded. Here N (Overall number of participants analyzed) signifies participants evaluable for this OM.
Measure: Mean (Standard Error); unit: Log10 copies*day per milliliter
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 483 | 1041
Log10 copies*day per milliliter | 823.7 (33.668) | 921.47 (25.706)

14. Secondary Outcome: Number of Participants With First Occurrence of Molecularly Confirmed Mild COVID-19 (Double Blind Phase
Description: Molecularly confirmed mild Covid-19 was defined as a SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (example, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample and one of the following signs and symptoms: fever (>=38°C or >=100.4°F), sore throat, malaise (loss of appetite, generally unwell, fatigue, physical weakness), headache, muscle pain (myalgia), gastrointestinal symptoms, cough, chest congestion, runny nose, wheezing, skin rash, eye irritation or discharge, chills, new or changing olfactory or taste disorders, red or bruised looking feet or toes, or shaking chills or rigors.
Time Frame: 14 Days after double-blind vaccination on Day1 (Day 15)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19400 | 19398
Participants | 11 | 15

15. Secondary Outcome: Number of Participants With First Occurrence of Molecularly Confirmed Mild COVID-19 (Double Blind Phase)
Description: as for outcome 14
Time Frame: 28 Days after double-blind vaccination on Day 1 (Day 29)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19113 | 18924
Participants | 10 | 12

16. Secondary Outcome: Number of Participants With First Occurrence of Molecularly Confirmed COVID-19 Defined by the US Food and Drug Administration (FDA) Harmonized Case Definition (Double Blind Phase)
Description: Molecularly confirmed COVID-19 was defined as a positive SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (example, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample; and COVID-19 symptoms consistent with those defined by the US FDA harmonized case definition at the time of finalization of the study protocol: fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, diarrhea.
Time Frame: 14 Days after double-blind vaccination on Day 1 (Day 15)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19400 | 19398
Participants | 492 | 1067

17. Secondary Outcome: Number of Participants With First Occurrence of Molecularly Confirmed COVID-19 Defined by the US Food and Drug Administration (FDA) Harmonized Case Definition (Double Blind Phase)
Description: as for outcome 16
Time Frame: 28 Days after double-blind vaccination on Day 1 (Day 29)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19113 | 18924
Participants | 441 | 884

18. Secondary Outcome: Number of Participants With Burden of Disease (BOD) Based on First Occurrence of Molecularly Confirmed Symptomatic COVID-19 (Double Blind Phase)
Description: BOD is a weighted version of the mild, moderate, and severe/critical vaccine efficacies and was evaluated based on the first occurrence of molecularly confirmed COVID-19, including mild, moderate or severe/critical COVID-19 case.
Time Frame: 14 Days after double-blind vaccination on Day 1 (Day 15)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19400 | 19398
Participants | 495 | 1082

19. Secondary Outcome: Number of Participants With BOD Based on First Occurrence of Molecularly Confirmed Symptomatic COVID-19 (Double Blind Phase)
Description: as for outcome 18
Time Frame: 28 Days after double-blind vaccination on Day 1 (Day 29)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19113 | 18924
Participants | 443 | 895

20. Secondary Outcome: Number of Participants With SARS-CoV-2 Seroconversion Based on Antibodies to N Protein Using ELISA and/or SARS-CoV-2 Immunoglobulin Assay (Double Blind Phase)
Description: Number of participants with SARS-CoV-2 seroconversion based on antibodies to nucleocapsid (N) protein using enzyme-linked immunosorbent assay (ELISA) and/or SARS-CoV- 2 immunoglobulin assay that is dependent on the SARS-CoV-2 N protein was reported.
Time Frame: From Day 29 until end of double-blind phase at Month 6
Population: PP set included participants of the FAS who received double-blind study vaccine and who were seronegative at the time of double-blind vaccination and who had no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine. Participants who had a COVID-19 case with an onset or discontinued before day 29 in PP set were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19113 | 18924
Participants | 550 | 724

21. Secondary Outcome: Number of Participants With Asymptomatic Infection Detected by RT-PCR at the Time of the Month 6/Unblinding Visit (Double Blind Phase)
Description: Number of participants with asymptomatic infection detected by RT-PCR at the time of the Month 6/unblinding visit were reported.
Time Frame: Month 6
Population: PP set included participants of the FAS who received double-blind study vaccine and who were seronegative at the time of double-blind vaccination and who had no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19113 | 18924
Participants | 10 | 12

22. Secondary Outcome: Number of Participants With First Occurrence of SARS-CoV-2 Infection (Serologically and/or Molecularly Confirmed) (Double Blind Phase)
Description: Number of participants with first occurrence of SARS-CoV-2 infection (serologically and/or molecularly confirmed) were reported.
Time Frame: 28 days after double-blind vaccination on Day 1 (Day 29)
Population: PP set included participants of the FAS who received double-blind study vaccine and who were seronegative at the time of double-blind vaccination and who had no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine. Here "N" signifies the excluded participants who had a COVID-19 case with an onset or discontinued before Day 29.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 19113 | 18924
Participants | 1038 | 1699

23. Secondary Outcome: Number of Participants With First Occurrence of Molecularly Confirmed, Moderate to Severe/Critical COVID-19 for Seronegative Participants (Double Blind Phase)
Description: Molecularly confirmed moderate to severe/critical COVID-19 was defined as a SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (example, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample. Moderate included one sign or symptom such as respiratory rate >= 20 breaths per minute and symptoms such as shortness of breath or two signs or symptoms such as heart rate >= 90 beats per minute (beats/minute) and symptoms such as cough from a list of signs and symptoms and severe/critical included one of the following signs and symptoms: respiratory rate >=30 breaths/minute, heart rate >=125 beats/minute,SpO2 <=93% on room air at sea level respiratory failure, evidence of shock, significant acute renal, hepatic, or neurologic dysfunction, admission to the ICU, death defined as per FDA guidance. Seronegative is defined as N-serology seronegative at the time of boosting or at the Year 1 visit if not boosted.
Time Frame: 1 day after double-blind vaccination on Day 1 (Day 2)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 21898 | 21890
Participants | 575 | 1189

24. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) (Double Blind Phase)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. SAE is any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Baseline (Day 1) up to 35 weeks
Population: FAS included all randomized participants with a documented double-blind study vaccine administration, regardless of the occurrence of protocol deviations and serostatus at enrollment. Here N (Overall number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 21894 | 21882
Participants | 235 | 358

25. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI) (Double Blind Phase)
Description: Number of participants with AESIs were reported. AESIs are significant AEs that are judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. Thrombosis with Thrombocytopenia Syndrome (TTS), a syndrome characterized by a combination of both a thrombotic event and thrombocytopenia, is considered to be an AESI in this study. A suspected TTS case is defined as: Thrombotic events: suspected deep vessel venous or arterial thrombotic events; Thrombocytopenia, defined as platelet count below 150,000/micro liter.
Time Frame: Baseline (Day 1) up to 35 weeks
Population: FAS included all randomized participants with a documented double-blind study vaccine administration, regardless of the occurrence of protocol deviations and serostatus at enrollment. Here N (Overall number of participants analyzed) signifies participants evaluated for this outcome measure (OM).
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 21894 | 21882
Participants | 6 | 5

26. Secondary Outcome: Number of Participants With Medically-Attended Adverse Events (MAAEs) (Double Blind Phase)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. MAAEs were defined as AEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason.
Time Frame: Up to 6 months after double-blind vaccination on Day 1 (up to 6 months)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 21894 | 21882
Participants | 1672 | 1885

27. Secondary Outcome: Number of Participants With MAAEs Leading to Study Discontinuation (Double Blind Phase)
Description: MAAEs were defined as AEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. Routine study visits were not considered medically-attended visits. New onset of chronic diseases was collected as part of the MAAEs.
Time Frame: Up to 35 weeks
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 21894 | 21882
Participants | 1 | 2

28. Secondary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) During 7 Days Following Vaccination (Double Blind Phase)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Participants who were enrolled in safety subset were asked to note in the e-Diary occurrences of injection site pain/tenderness, erythema, and swelling at the study vaccine injection site daily for 7 days post-vaccination (day of vaccination and the subsequent 7 days).
Time Frame: Up to Day 8 (7 Days after double-blind vaccination on Day 1)
Population: Safety population is a subset of FAS for the analysis of solicited local adverse event. Here N (Overall number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 3356 | 3379
Participants | 1839 | 684

29. Secondary Outcome: Number of Participants With Solicited Systemic AEs During 7 Days Following Vaccination (Double Blind Phase)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with pharmaceutical/biological agent under study. Participants who were enrolled in safety subset were instructed on how to record daily temperature using a thermometer provided for home use. Participants recorded the temperature in the e-Diary in the evening of the day of vaccination, and then daily for the next 7 days approximately at the same time each day. If more than 1 measurement was made on any given day, the highest temperature of that day was recorded in the e-Diary. Fever was defined as endogenous elevation of body temperature >= 38.0 degree Celsius or >=100.4-degree Fahrenheit, as recorded in at least 1 measurement. Participants also noted the signs and symptoms in the e-Diary on a daily basis for 7 days post vaccination (day of vaccination and the subsequent 7 days), for the following events: fatigue, headache, nausea, myalgia.
Time Frame: Up to Day 8 (7 Days after double-blind vaccination on Day 1)
Population: Safety population is a subset of FAS for the analysis of solicited systemic adverse event. Here N (Overall number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 3356 | 3379
Participants | 2021 | 1307

30. Secondary Outcome: Number of Participants With Unsolicited AEs During 28 Days Post-vaccination (Double Blind Phase)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: Up to Day 29 (28 Days after double-blind vaccination on Day 1)
Population: Safety population is a subset of FAS for the analysis of unsolicited adverse event. Here N (Overall number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 3356 | 3379
Participants | 456 | 422

31. Secondary Outcome: Binding Antibodies to SARS-CoV-2 S Protein Assessed by ELISA (Double Blind Phase)
Description: Binding antibodies to SARS-CoV-2 S protein as assessed by enzyme-linked immunosorbent assay (ELISA) to measure humoral immune response was reported. The lower limit of quantification (LLOQ) and upper limit of quantification (ULOQ) were 50.3 EU/mL and 58,158.10 EU/mL, respectively. A sample was considered positive if the value was strictly greater than the LLOQ (>LLOQ).
Time Frame: Baseline (Day 1), Day 29, and Day 71
Population: PPI set included all randomized and vaccinated participants, including those who were part of the immunogenicity subset and for whom immunogenicity data were available, excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. Here N (Overall number of participants analyzed) signifies participants evaluated for this outcome measure and 'n' (number analyzed) signifies number of participants evaluable at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per milliliter (EU/mL)
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo
Number analyzed (Participants) | 193 | 167
ELISA units per milliliter (EU/mL)
  Baseline (Day 1) | NA [NA to NA] — Here NA signifies that the sample was not positive as Geometric mean, and 95% confidence interval value were less than LLOQ i.e., 50.3 EU/mL. | NA [NA to NA] — Here NA signifies that the sample was not positive as Geometric mean, and 95% confidence interval value were less than LLOQ i.e., 50.3 EU/mL.
  Day 29: number analyzed (Participants) | 177 | 154
  Day 29 | 336 [284 to 398] | NA [NA to NA] — Here NA signifies that the sample was not positive as Geometric mean, and 95% confidence interval value were less than LLOQ i.e., 50.3 EU/mL.
  Day 71: number analyzed (Participants) | 164 | 138
  Day 71 | 526 [437 to 633] | NA [NA to NA] — Here NA signifies that the sample was not positive as Geometric mean, and 95% confidence interval value were less than LLOQ i.e., 50.3 EU/mL.

32. Secondary Outcome: Number of Participants With Antibody Titers to Ad26.COV2.S (Booster Phase)
Description: Number of participants with antibody titers to Ad26.COV2.S to measure immune response were reported.
Time Frame: 28 days after booster vaccination on Day 365 (up to Day 393)
Population: PPI booster analysis set included all participants who received an Ad26.COV2.S booster dose (Year 1(Week 52)/Booster Visit) and who had been selected for inclusion in homologous or heterologous booster subset as of protocol amendment 6. This OM was planned to be analyzed based on homologous and heterologous booster groups. Here, "0" participants in "overall number of participants analyzed" field indicated that data for this OM was not collected and analyzed due to change in planned analysis.
Groups:
- Homologous Booster Group (2 Doses of Ad26.COV2.S 5*10^10 vp): As per protocol amendment 6, in homologous booster group participants received 2 doses of Ad26.COV2.S 5*10^10 vp (Ad26.COV2.S booster vaccination following an early or late first Ad26.COV2.S vaccination) as early booster group in which duration between the 2 doses of Ad26.COV2.S 5*10^10 vp was less than (<) 6 months or late booster group in which duration between the 2 doses of Ad26.COV2.S. was >=6 months.
- Heterologous Booster Group: Placebo + 2 Doses of mRNA Vaccine + Ad26.COV2.S 5*10^10 vp: As per protocol amendment 6, participants who received placebo at Day 1 during the double blind phase and had received primary vaccination with an mRNA vaccine outside of the study further received Ad26.COV2.S 5*10^10 vp booster vaccination at Year 1 booster visit.
- Heterologous Booster Group: Ad26.COV2.S 5*10^10 vp Booster After Any Other Schedule: As per protocol amendment 6, participants who received placebo on Day 1 in the double-blind phase and had received primary vaccination with any other COVID-19 vaccination schedule outside of the study that is other adenoviral vector, further received an Ad26.COV2.S 5*10^10 vp booster vaccination at Year 1 booster vaccination visit.
- Heterologous Booster Group: Inactivated Vaccine + Ad26.COV2.S 5*10^10 vp: As per protocol amendment 6, participants who received placebo in the double-blind phase and had received primary vaccination with inactivated vaccine further received an Ad26.COV2.S 5*10^10 vp booster vaccination at Year 1 booster vaccination visit.
Arm/Group | Homologous Booster Group (2 Doses of Ad26.COV2.S 5*10^10 vp) | Heterologous Booster Group: Placebo + 2 Doses of mRNA Vaccine + Ad26.COV2.S 5*10^10 vp | Heterologous Booster Group: Ad26.COV2.S 5*10^10 vp Booster After Any Other Schedule | Heterologous Booster Group: Inactivated Vaccine + Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 0 | 0 | 0 | 0

33. Secondary Outcome: Number of Participants With Binding Antibodies to SARS- CoV-2S Protein as Measured by ELISA (Booster Phase)
Description: Number of participants with binding antibodies to SARS- CoV-2S protein as measured by ELISA was reported.
Time Frame: 29 days after booster vaccination on Day 365 (Day 394)
Population: Per protocol booster immunogenicity analysis set included all participants who received an Ad26.COV2.S booster dose (Year 1 [Week 52]/Booster Visit) and who had been selected for inclusion in the homologous or heterologous booster subset as of protocol amendment 6. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure. As planned, this outcome measure was analyzed based on homologous and heterologous booster groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Homologous Booster Group (2 Doses of Ad26.COV2.S 5*10^10 vp) | Heterologous Booster Group: Placebo + 2 Doses of mRNA Vaccine + Ad26.COV2.S 5*10^10 vp | Heterologous Booster Group: Ad26.COV2.S 5*10^10 vp Booster After Any Other Schedule | Heterologous Booster Group: Inactivated Vaccine + Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 88 | 29 | 25 | 11
Participants | 64 | 26 | 9 | 3

ADVERSE EVENTS:
Time Frame: DB phase: All-cause mortality and SAEs: Baseline (Day 1) up to 35 weeks; Other AEs: Day 1 till 28 days after first vaccination; All participants Arm: all-cause mortality and SAEs: Day 1 up to end of study (up to 2 years 6.5 months); Booster treatment groups: Other AEs: from Day 1 till 28 days after booster vaccination on Day 365 (up to Day 393). Solicited AEs: 7 days after first/booster vaccination
Description: Per change in planned analysis: data for DB & OL phase (booster arms) was collected & reported in 'All participants' arms for all-cause mortality and SAEs. Thus, at risk=0 for booster arms. Other AEs: per plan, Safety subset (subset of FAS) was used and hence at risk=0 for 'All participants' arm as this arm had all treated participants. AEs in DB arms were coded with MedDRA Version 24.0. Same AEs might differ in names in both phases due to coding with different MedDRA versions.
Arm/Group | Double-blind Phase: Ad26.COV2.S 5*10^10 vp | Double-blind Phase: Placebo | Combined Double-blind and Open-label Phase: All Participants | OL Phase: Ad26.COV2.S 5*10^10 vp + Ad26.COV2.S 5*10^10 vp Booster | Open Label Phase: mRNA 2 Dose Schedule + Ad26.COV2.S 5*10^10 vp Booster | OL Phase: Non-mRNA Any Schedule +Ad26.COV2.S vp Booster OR mRNA Other Schedule +Ad26.COV2.S Booster
All-Cause Mortality (participants affected / at risk) | 36/21898 | 64/21890 | 324/43788 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 235/21898 | 358/21890 | 2758/43788 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 2451/3356 | 1653/3380 | 0/0 | 6048/22213 | 190/613 | 315/943
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase: Ad26.COV2.S 5*10^10 vp (N=21898) | Double-blind Phase: Placebo (N=21890) | Combined Double-blind and Open-label Phase: All Participants (N=43788) | OL Phase: Ad26.COV2.S 5*10^10 vp + Ad26.COV2.S 5*10^10 vp Booster (N=0) | Open Label Phase: mRNA 2 Dose Schedule + Ad26.COV2.S 5*10^10 vp Booster (N=0) | OL Phase: Non-mRNA Any Schedule +Ad26.COV2.S vp Booster OR mRNA Other Schedule +Ad26.COV2.S Booster (N=0)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 18 | NA | NA | NA
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 1 | NA | NA | NA
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 0 | 1 | NA | NA | NA
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 6 | NA | NA | NA
Elephantiasis (Blood and lymphatic system disorders) | 0 | 0 | 1 | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | NA | NA | NA
Granulomatous lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | NA | NA | NA
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | NA | NA | NA
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | NA | NA | NA
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 3 | 13 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | NA | NA | NA
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2 | NA | NA | NA
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | NA | NA | NA
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | NA | NA | NA
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | NA | NA | NA
Splenic thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | NA | NA | NA
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 0 | 1 | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 24 | NA | NA | NA
Acute cardiac event (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Acute coronary syndrome (Cardiac disorders) | 0 | 2 | 14 | NA | NA | NA
Acute myocardial infarction (Cardiac disorders) | 2 | 7 | 53 | NA | NA | NA
Angina pectoris (Cardiac disorders) | 0 | 1 | 7 | NA | NA | NA
Angina unstable (Cardiac disorders) | 0 | 0 | 10 | NA | NA | NA
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 1 | NA | NA | NA
Arrhythmia (Cardiac disorders) | 0 | 2 | 9 | NA | NA | NA
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 2 | NA | NA | NA
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 1 | 6 | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 47 | NA | NA | NA
Atrial flutter (Cardiac disorders) | 0 | 2 | 5 | NA | NA | NA
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 3 | NA | NA | NA
Atrioventricular block (Cardiac disorders) | 0 | 0 | 2 | NA | NA | NA
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 3 | NA | NA | NA
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Atrioventricular node dysfunction (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Bradycardia (Cardiac disorders) | 0 | 0 | 6 | NA | NA | NA
Cardiac amyloidosis (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Cardiac arrest (Cardiac disorders) | 0 | 2 | 12 | NA | NA | NA
Cardiac disorder (Cardiac disorders) | 0 | 1 | 1 | NA | NA | NA
Cardiac failure (Cardiac disorders) | 2 | 4 | 19 | NA | NA | NA
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 5 | NA | NA | NA
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Cardiac failure congestive (Cardiac disorders) | 2 | 4 | 16 | NA | NA | NA
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 0 | 2 | NA | NA | NA
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 5 | NA | NA | NA
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Chronic left ventricular failure (Cardiac disorders) | 0 | 0 | 2 | NA | NA | NA
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 2 | NA | NA | NA
Cor pulmonale (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Coronary artery disease (Cardiac disorders) | 2 | 0 | 35 | NA | NA | NA
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 3 | NA | NA | NA
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 1 | NA | NA | NA
Coronary artery thrombosis (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Mitral valve disease (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 3 | NA | NA | NA
Mitral valve prolapse (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Mitral valve stenosis (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Myocardial infarction (Cardiac disorders) | 2 | 3 | 23 | NA | NA | NA
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 8 | NA | NA | NA
Myocarditis (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Palpitations (Cardiac disorders) | 0 | 0 | 2 | NA | NA | NA
Pericarditis (Cardiac disorders) | 1 | 0 | 2 | NA | NA | NA
Pericarditis constrictive (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2 | NA | NA | NA
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 2 | NA | NA | NA
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 4 | NA | NA | NA
Tachycardia (Cardiac disorders) | 0 | 1 | 2 | NA | NA | NA
Tachycardia paroxysmal (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 2 | NA | NA | NA
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 2 | NA | NA | NA
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 0 | 1 | NA | NA | NA
Pseudoxanthoma elasticum (Congenital, familial and genetic disorders) | 0 | 0 | 1 | NA | NA | NA
Rathke's cleft cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1 | NA | NA | NA
Skeletal dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | NA | NA | NA
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 2 | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 5 | NA | NA | NA
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 3 | NA | NA | NA
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | NA | NA | NA
Basedow's disease (Endocrine disorders) | 0 | 0 | 1 | NA | NA | NA
Endocrine disorder (Endocrine disorders) | 0 | 0 | 1 | NA | NA | NA
Goitre (Endocrine disorders) | 0 | 0 | 2 | NA | NA | NA
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 1 | NA | NA | NA
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 0 | 1 | NA | NA | NA
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | NA | NA | NA
Thyroid mass (Endocrine disorders) | 0 | 0 | 3 | NA | NA | NA
Blindness (Eye disorders) | 0 | 0 | 1 | NA | NA | NA
Cataract (Eye disorders) | 0 | 0 | 2 | NA | NA | NA
Diplopia (Eye disorders) | 1 | 2 | 4 | NA | NA | NA
Endocrine ophthalmopathy (Eye disorders) | 0 | 0 | 1 | NA | NA | NA
Glaucoma (Eye disorders) | 0 | 0 | 1 | NA | NA | NA
Macular degeneration (Eye disorders) | 0 | 0 | 1 | NA | NA | NA
Retinal artery embolism (Eye disorders) | 0 | 0 | 1 | NA | NA | NA
Retinal detachment (Eye disorders) | 0 | 0 | 3 | NA | NA | NA
Retinal vascular thrombosis (Eye disorders) | 0 | 0 | 1 | NA | NA | NA
Retinal vein thrombosis (Eye disorders) | 1 | 0 | 1 | NA | NA | NA
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1 | NA | NA | NA
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 7 | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 6 | NA | NA | NA
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Abdominal wall disorder (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 2 | NA | NA | NA
Anal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Colitis (Gastrointestinal disorders) | 1 | 1 | 3 | NA | NA | NA
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 2 | NA | NA | NA
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1 | 1 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | NA | NA | NA
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Enteritis (Gastrointestinal disorders) | 1 | 0 | 4 | NA | NA | NA
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Epiploic appendagitis (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Gallstone ileus (Gastrointestinal disorders) | 0 | 1 | 1 | NA | NA | NA
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 4 | NA | NA | NA
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 4 | NA | NA | NA
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Gastritis (Gastrointestinal disorders) | 0 | 0 | 4 | NA | NA | NA
Gastritis alcoholic (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 10 | NA | NA | NA
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | NA | NA | NA
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Gastrointestinal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 3 | NA | NA | NA
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 3 | NA | NA | NA
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 4 | NA | NA | NA
Hernial eventration (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 7 | NA | NA | NA
Hiatus hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Ileus (Gastrointestinal disorders) | 0 | 0 | 3 | NA | NA | NA
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 2 | NA | NA | NA
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 14 | NA | NA | NA
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Internal hernia (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Intestinal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 3 | NA | NA | NA
Intestinal mass (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 2 | 3 | 23 | NA | NA | NA
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 3 | NA | NA | NA
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 1 | NA | NA | NA
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Lumbar hernia (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Melaena (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Mesenteric panniculitis (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1 | NA | NA | NA
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 12 | NA | NA | NA
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 5 | NA | NA | NA
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 4 | NA | NA | NA
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | NA | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 3 | 16 | NA | NA | NA
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 3 | NA | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 10 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | NA | NA | NA
Accidental death (General disorders) | 1 | 0 | 5 | NA | NA | NA
Asthenia (General disorders) | 0 | 0 | 1 | NA | NA | NA
Chest pain (General disorders) | 3 | 2 | 23 | NA | NA | NA
Complication associated with device (General disorders) | 0 | 0 | 1 | NA | NA | NA
Cyst (General disorders) | 0 | 0 | 1 | NA | NA | NA
Death (General disorders) | 7 | 4 | 59 | NA | NA | NA
Drowning (General disorders) | 1 | 0 | 3 | NA | NA | NA
Drug withdrawal syndrome (General disorders) | 1 | 0 | 3 | NA | NA | NA
Fatigue (General disorders) | 0 | 0 | 1 | NA | NA | NA
Gait disturbance (General disorders) | 0 | 1 | 2 | NA | NA | NA
Generalised oedema (General disorders) | 0 | 0 | 1 | NA | NA | NA
Illness (General disorders) | 0 | 0 | 1 | NA | NA | NA
Implant site inflammation (General disorders) | 0 | 0 | 1 | NA | NA | NA
Malaise (General disorders) | 0 | 1 | 1 | NA | NA | NA
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 4 | NA | NA | NA
Non-cardiac chest pain (General disorders) | 0 | 0 | 4 | NA | NA | NA
Oedema peripheral (General disorders) | 2 | 0 | 4 | NA | NA | NA
Pain (General disorders) | 0 | 0 | 1 | NA | NA | NA
Pelvic mass (General disorders) | 0 | 0 | 2 | NA | NA | NA
Procedural failure (General disorders) | 0 | 0 | 1 | NA | NA | NA
Pyrexia (General disorders) | 1 | 1 | 5 | NA | NA | NA
Stent-graft endoleak (General disorders) | 0 | 0 | 1 | NA | NA | NA
Sudden cardiac death (General disorders) | 0 | 0 | 3 | NA | NA | NA
Sudden death (General disorders) | 1 | 3 | 10 | NA | NA | NA
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1 | NA | NA | NA
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 5 | NA | NA | NA
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Biliary tract disorder (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 2 | NA | NA | NA
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Cholecystitis (Hepatobiliary disorders) | 3 | 1 | 18 | NA | NA | NA
Cholecystitis acute (Hepatobiliary disorders) | 2 | 1 | 19 | NA | NA | NA
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 2 | NA | NA | NA
Cholecystocholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 32 | NA | NA | NA
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 2 | NA | NA | NA
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 4 | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 2 | NA | NA | NA
ABO incompatibility (Immune system disorders) | 0 | 0 | 1 | NA | NA | NA
Allergy to chemicals (Immune system disorders) | 0 | 1 | 1 | NA | NA | NA
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 6 | NA | NA | NA
Anaphylactic shock (Immune system disorders) | 0 | 0 | 2 | NA | NA | NA
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | NA | NA | NA
Hypersensitivity (Immune system disorders) | 1 | 0 | 1 | NA | NA | NA
Sarcoidosis (Immune system disorders) | 0 | 0 | 2 | NA | NA | NA
Abdominal sepsis (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Abscess (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Abscess limb (Infections and infestations) | 1 | 2 | 4 | NA | NA | NA
Abscess neck (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Abscess soft tissue (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Acute hepatitis B (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Anal abscess (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Appendicitis (Infections and infestations) | 10 | 8 | 54 | NA | NA | NA
Appendicitis perforated (Infections and infestations) | 1 | 0 | 3 | NA | NA | NA
Arthritis bacterial (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Arthritis gonococcal (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Arthritis infective (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Bacteraemia (Infections and infestations) | 0 | 1 | 2 | NA | NA | NA
Bacterial diarrhoea (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Bacterial food poisoning (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Bacterial infection (Infections and infestations) | 0 | 1 | 2 | NA | NA | NA
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Biliary sepsis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Biliary tract infection (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Brain abscess (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Bronchitis (Infections and infestations) | 0 | 0 | 4 | NA | NA | NA
Bullous erysipelas (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Bursitis infective (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
COVID-19 (Infections and infestations) | 5 | 53 | 146 | NA | NA | NA
COVID-19 pneumonia (Infections and infestations) | 9 | 45 | 105 | NA | NA | NA
Campylobacter infection (Infections and infestations) | 1 | 0 | 2 | NA | NA | NA
Cardiac valve abscess (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Cavernous sinus thrombosis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Cellulitis (Infections and infestations) | 2 | 2 | 23 | NA | NA | NA
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Chronic sinusitis (Infections and infestations) | 0 | 1 | 2 | NA | NA | NA
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 2 | NA | NA | NA
Colonic abscess (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Complicated appendicitis (Infections and infestations) | 0 | 1 | 3 | NA | NA | NA
Creutzfeldt-Jakob disease (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Cystitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 2 | NA | NA | NA
Dengue fever (Infections and infestations) | 0 | 0 | 4 | NA | NA | NA
Dengue haemorrhagic fever (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Diabetic foot infection (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Diverticulitis (Infections and infestations) | 1 | 0 | 15 | NA | NA | NA
Diverticulitis intestinal perforated (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Dysentery (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Encephalitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Endocarditis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Epiglottitis (Infections and infestations) | 1 | 0 | 1 | NA | NA | NA
Epstein-Barr virus infection (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Escherichia infection (Infections and infestations) | 1 | 0 | 1 | NA | NA | NA
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Eye abscess (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Focal peritonitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Gangrene (Infections and infestations) | 0 | 1 | 3 | NA | NA | NA
Gastroenteritis (Infections and infestations) | 3 | 2 | 17 | NA | NA | NA
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Genital abscess (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
HIV infection (Infections and infestations) | 0 | 0 | 6 | NA | NA | NA
Hepatitis B (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Herpes zoster meningitis (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Implant site infection (Infections and infestations) | 1 | 0 | 1 | NA | NA | NA
Infected bite (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Infection (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Influenza (Infections and infestations) | 0 | 1 | 4 | NA | NA | NA
Labyrinthitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Large intestine infection (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Laryngitis (Infections and infestations) | 1 | 0 | 1 | NA | NA | NA
Liver abscess (Infections and infestations) | 1 | 0 | 3 | NA | NA | NA
Lower respiratory tract infection (Infections and infestations) | 1 | 3 | 11 | NA | NA | NA
Lung abscess (Infections and infestations) | 1 | 0 | 1 | NA | NA | NA
Mastoiditis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Medical device site infection (Infections and infestations) | 1 | 0 | 1 | NA | NA | NA
Meningitis (Infections and infestations) | 1 | 0 | 3 | NA | NA | NA
Meningitis bacterial (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Meningitis cryptococcal (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Meningitis tuberculous (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Monkeypox (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Mononucleosis syndrome (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Neurosyphilis (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Orchitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Osteomyelitis (Infections and infestations) | 1 | 1 | 16 | NA | NA | NA
Pelvic abscess (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Perichondritis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Perineal abscess (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 1 | NA | NA | NA
Perirectal abscess (Infections and infestations) | 1 | 0 | 1 | NA | NA | NA
Peritoneal abscess (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Peritonitis (Infections and infestations) | 0 | 0 | 3 | NA | NA | NA
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 2 | NA | NA | NA
Pertussis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Pilonidal disease (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Plasmodium vivax infection (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 3 | NA | NA | NA
Pneumonia (Infections and infestations) | 8 | 13 | 56 | NA | NA | NA
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 7 | NA | NA | NA
Pneumonia bacterial (Infections and infestations) | 0 | 2 | 18 | NA | NA | NA
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Pneumonia viral (Infections and infestations) | 2 | 1 | 2 | NA | NA | NA
Post procedural infection (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Post procedural sepsis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Postoperative wound infection (Infections and infestations) | 0 | 0 | 5 | NA | NA | NA
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Psoas abscess (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Pulmonary tuberculosis (Infections and infestations) | 2 | 1 | 8 | NA | NA | NA
Pyelonephritis (Infections and infestations) | 1 | 0 | 7 | NA | NA | NA
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Rectal abscess (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Renal abscess (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 1 | NA | NA | NA
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Scrotal abscess (Infections and infestations) | 1 | 0 | 1 | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 2 | 22 | NA | NA | NA
Septic shock (Infections and infestations) | 0 | 0 | 10 | NA | NA | NA
Severe acute respiratory syndrome (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Soft tissue infection (Infections and infestations) | 1 | 0 | 4 | NA | NA | NA
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 2 | NA | NA | NA
Staphylococcal osteomyelitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Subdiaphragmatic abscess (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Suspected COVID-19 (Infections and infestations) | 0 | 1 | 2 | NA | NA | NA
Thyroglossal cyst infection (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Tonsillitis (Infections and infestations) | 1 | 0 | 2 | NA | NA | NA
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Tuberculosis (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Typhoid fever (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 3 | NA | NA | NA
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Urinary tract candidiasis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 4 | 3 | 32 | NA | NA | NA
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 4 | NA | NA | NA
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Urosepsis (Infections and infestations) | 0 | 0 | 10 | NA | NA | NA
Viral infection (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Wound infection (Infections and infestations) | 0 | 1 | 3 | NA | NA | NA
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 3 | NA | NA | NA
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 2 | NA | NA | NA
Anastomotic complication (Injury, poisoning and procedural complications) | 0 | 1 | 1 | NA | NA | NA
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1 | NA | NA | NA
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 14 | NA | NA | NA
Aortic injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 3 | NA | NA | NA
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 4 | NA | NA | NA
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 4 | NA | NA | NA
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 | 2 | 12 | NA | NA | NA
Exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 3 | NA | NA | NA
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 6 | NA | NA | NA
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1 | 20 | NA | NA | NA
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3 | NA | NA | NA
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 3 | NA | NA | NA
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | NA | NA | NA
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Gastrointestinal anastomotic complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 4 | NA | NA | NA
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1 | 7 | NA | NA | NA
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 7 | NA | NA | NA
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 11 | NA | NA | NA
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 1 | NA | NA | NA
Incision site impaired healing (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 2 | NA | NA | NA
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 3 | NA | NA | NA
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 3 | NA | NA | NA
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 4 | NA | NA | NA
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 2 | NA | NA | NA
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 5 | NA | NA | NA
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 2 | NA | NA | NA
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 1 | 7 | NA | NA | NA
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 7 | NA | NA | NA
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 5 | NA | NA | NA
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 4 | NA | NA | NA
Multiple injuries (Injury, poisoning and procedural complications) | 2 | 1 | 7 | NA | NA | NA
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | NA | NA | NA
Nasal injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | NA | NA | NA
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 3 | NA | NA | NA
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 3 | NA | NA | NA
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 6 | NA | NA | NA
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 3 | NA | NA | NA
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 4 | NA | NA | NA
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 3 | NA | NA | NA
Post procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Post vaccination syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 1 | NA | NA | NA
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | NA | NA | NA
Prescribed overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 9 | NA | NA | NA
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 7 | NA | NA | NA
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 5 | NA | NA | NA
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 2 | NA | NA | NA
Soft tissue foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Soft tissue injury (Injury, poisoning and procedural complications) | 2 | 1 | 8 | NA | NA | NA
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Splenic injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Stab wound (Injury, poisoning and procedural complications) | 0 | 1 | 5 | NA | NA | NA
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 4 | NA | NA | NA
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 8 | NA | NA | NA
Testicular injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 4 | NA | NA | NA
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 3 | 14 | NA | NA | NA
Tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | NA | NA | NA
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | NA | NA | NA
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 6 | NA | NA | NA
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 1 | NA | NA | NA
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 2 | NA | NA | NA
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 3 | NA | NA | NA
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 4 | NA | NA | NA
Arthroscopy (Investigations) | 0 | 0 | 1 | NA | NA | NA
Blood pressure increased (Investigations) | 0 | 0 | 1 | NA | NA | NA
Carcinoembryonic antigen increased (Investigations) | 0 | 0 | 1 | NA | NA | NA
HIV test positive (Investigations) | 1 | 0 | 1 | NA | NA | NA
Haemoglobin decreased (Investigations) | 0 | 1 | 3 | NA | NA | NA
Liver function test increased (Investigations) | 0 | 0 | 1 | NA | NA | NA
Micrococcus test positive (Investigations) | 0 | 0 | 1 | NA | NA | NA
Misleading laboratory test result (Investigations) | 0 | 0 | 1 | NA | NA | NA
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | NA | NA | NA
Oxygen saturation decreased (Investigations) | 0 | 0 | 1 | NA | NA | NA
Platelet count decreased (Investigations) | 0 | 0 | 5 | NA | NA | NA
Pulse absent (Investigations) | 0 | 1 | 1 | NA | NA | NA
SARS-CoV-2 test positive (Investigations) | 0 | 2 | 4 | NA | NA | NA
Thyroid function test abnormal (Investigations) | 0 | 0 | 1 | NA | NA | NA
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | NA | NA | NA
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 4 | NA | NA | NA
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 4 | NA | NA | NA
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 2 | 9 | NA | NA | NA
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0 | 1 | NA | NA | NA
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Histamine intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 5 | NA | NA | NA
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 8 | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 8 | NA | NA | NA
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 2 | NA | NA | NA
Obesity (Metabolism and nutrition disorders) | 2 | 0 | 17 | NA | NA | NA
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 6 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6 | NA | NA | NA
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | NA | NA | NA
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 11 | NA | NA | NA
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | NA | NA | NA
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | NA | NA | NA
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | NA | NA | NA
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Immunoglobulin G4 related disease (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | NA | NA | NA
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 17 | NA | NA | NA
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 10 | NA | NA | NA
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 54 | NA | NA | NA
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | NA | NA | NA
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | NA | NA | NA
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | NA | NA | NA
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 4 | 11 | NA | NA | NA
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | NA | NA | NA
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | NA | NA | NA
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | NA | NA | NA
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | NA | NA | NA
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | NA | NA | NA
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | NA | NA | NA
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 8 | NA | NA | NA
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Anal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 9 | NA | NA | NA
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 8 | NA | NA | NA
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Bladder squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | NA | NA | NA
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 32 | NA | NA | NA
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 6 | NA | NA | NA
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | NA | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | NA | NA | NA
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 5 | NA | NA | NA
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | NA | NA | NA
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 8 | NA | NA | NA
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | NA | NA | NA
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | NA | NA | NA
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 7 | NA | NA | NA
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 6 | NA | NA | NA
Ewing's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Follicular lymphoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Follicular lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | NA | NA | NA
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 4 | NA | NA | NA
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | NA | NA | NA
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Hepatobiliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 10 | NA | NA | NA
Intraosseous meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | NA | NA | NA
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 10 | NA | NA | NA
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | NA | NA | NA
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 12 | NA | NA | NA
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 7 | NA | NA | NA
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Lymphoplasmacytoid lymphoma/immunocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | NA | NA | NA
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Malignant melanoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | NA | NA | NA
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | NA | NA | NA
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Neoplasm of orbit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | NA | NA | NA
Neuroectodermal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Neuroendocrine carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | NA | NA | NA
Neurofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | NA | NA | NA
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 4 | NA | NA | NA
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Ovarian germ cell teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Ovarian granulosa cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 6 | NA | NA | NA
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | NA | NA | NA
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 8 | NA | NA | NA
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Peritoneal mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | NA | NA | NA
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4 | NA | NA | NA
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 38 | NA | NA | NA
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | NA | NA | NA
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 6 | NA | NA | NA
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | NA | NA | NA
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | NA | NA | NA
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | NA | NA | NA
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | NA | NA | NA
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 4 | NA | NA | NA
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | NA | NA | NA
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | NA | NA | NA
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | NA | NA | NA
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 13 | NA | NA | NA
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Apallic syndrome (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Ascending flaccid paralysis (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Bell's palsy (Nervous system disorders) | 2 | 0 | 8 | NA | NA | NA
Brain stem thrombosis (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Carotid artery aneurysm (Nervous system disorders) | 0 | 0 | 3 | NA | NA | NA
Carotid artery disease (Nervous system disorders) | 0 | 0 | 2 | NA | NA | NA
Carotid artery dissection (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Carotid artery occlusion (Nervous system disorders) | 0 | 1 | 1 | NA | NA | NA
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 1 | NA | NA | NA
Cerebral haemorrhage (Nervous system disorders) | 1 | 1 | 5 | NA | NA | NA
Cerebral infarction (Nervous system disorders) | 1 | 2 | 4 | NA | NA | NA
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 8 | NA | NA | NA
Cerebral vasoconstriction (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 | 1 | 2 | NA | NA | NA
Cerebrospinal fistula (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 2 | NA | NA | NA
Cerebrovascular accident (Nervous system disorders) | 3 | 6 | 19 | NA | NA | NA
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 2 | NA | NA | NA
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Coma (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Complex regional pain syndrome (Nervous system disorders) | 1 | 0 | 1 | NA | NA | NA
Dizziness (Nervous system disorders) | 0 | 1 | 4 | NA | NA | NA
Embolic stroke (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Encephalopathy (Nervous system disorders) | 0 | 0 | 2 | NA | NA | NA
Epilepsy (Nervous system disorders) | 0 | 2 | 5 | NA | NA | NA
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 3 | NA | NA | NA
Guillain-Barre syndrome (Nervous system disorders) | 1 | 1 | 6 | NA | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 2 | NA | NA | NA
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 4 | NA | NA | NA
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Headache (Nervous system disorders) | 0 | 0 | 9 | NA | NA | NA
Hemiparesis (Nervous system disorders) | 2 | 0 | 5 | NA | NA | NA
Hemiplegia (Nervous system disorders) | 0 | 1 | 1 | NA | NA | NA
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 2 | NA | NA | NA
Hydrocephalus (Nervous system disorders) | 1 | 0 | 3 | NA | NA | NA
Hyperglycaemic seizure (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1 | 1 | NA | NA | NA
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Idiopathic intracranial hypertension (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Intracranial aneurysm (Nervous system disorders) | 1 | 1 | 5 | NA | NA | NA
Intracranial mass (Nervous system disorders) | 1 | 0 | 2 | NA | NA | NA
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 2 | NA | NA | NA
Ischaemic stroke (Nervous system disorders) | 3 | 0 | 45 | NA | NA | NA
Lacunar stroke (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 6 | NA | NA | NA
Metabolic encephalopathy (Nervous system disorders) | 1 | 1 | 3 | NA | NA | NA
Migraine (Nervous system disorders) | 0 | 1 | 5 | NA | NA | NA
Migraine without aura (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 2 | NA | NA | NA
Myelopathy (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Neuralgic amyotrophy (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Neuroglycopenia (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Optic neuritis (Nervous system disorders) | 0 | 1 | 2 | NA | NA | NA
Paraparesis (Nervous system disorders) | 0 | 1 | 1 | NA | NA | NA
Partial seizures (Nervous system disorders) | 0 | 0 | 3 | NA | NA | NA
Presyncope (Nervous system disorders) | 0 | 0 | 2 | NA | NA | NA
Radiculopathy (Nervous system disorders) | 0 | 0 | 3 | NA | NA | NA
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Sciatica (Nervous system disorders) | 0 | 0 | 5 | NA | NA | NA
Seizure (Nervous system disorders) | 1 | 0 | 15 | NA | NA | NA
Spinal cord compression (Nervous system disorders) | 0 | 1 | 1 | NA | NA | NA
Spinal cord haematoma (Nervous system disorders) | 0 | 1 | 1 | NA | NA | NA
Spondylitic myelopathy (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 5 | NA | NA | NA
Syncope (Nervous system disorders) | 2 | 2 | 28 | NA | NA | NA
Tension headache (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Transient global amnesia (Nervous system disorders) | 1 | 0 | 4 | NA | NA | NA
Transient ischaemic attack (Nervous system disorders) | 1 | 3 | 27 | NA | NA | NA
Transverse sinus thrombosis (Nervous system disorders) | 1 | 0 | 1 | NA | NA | NA
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Uraemic encephalopathy (Nervous system disorders) | 0 | 1 | 1 | NA | NA | NA
Vertebrobasilar artery dissection (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 4 | NA | NA | NA
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 4 | NA | NA | NA
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | NA | NA | NA
Abortion of ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | NA | NA | NA
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 21 | NA | NA | NA
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | NA | NA | NA
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 5 | NA | NA | NA
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | NA | NA | NA
Foetal growth abnormality (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | NA | NA | NA
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | NA | NA | NA
High risk pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | NA | NA | NA
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | NA | NA | NA
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | NA | NA | NA
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | NA | NA | NA
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | NA | NA | NA
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | NA | NA | NA
Vanishing twin syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | NA | NA | NA
Device breakage (Product Issues) | 0 | 0 | 2 | NA | NA | NA
Device dislocation (Product Issues) | 0 | 0 | 2 | NA | NA | NA
Device failure (Product Issues) | 0 | 0 | 1 | NA | NA | NA
Device power source issue (Product Issues) | 0 | 0 | 1 | NA | NA | NA
Drug delivery system malfunction (Product Issues) | 0 | 0 | 1 | NA | NA | NA
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 3 | NA | NA | NA
Anxiety (Psychiatric disorders) | 1 | 1 | 6 | NA | NA | NA
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 5 | NA | NA | NA
Borderline personality disorder (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Catatonia (Psychiatric disorders) | 1 | 0 | 1 | NA | NA | NA
Completed suicide (Psychiatric disorders) | 0 | 2 | 7 | NA | NA | NA
Confusional state (Psychiatric disorders) | 0 | 0 | 3 | NA | NA | NA
Conversion disorder (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Delirium (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Depression (Psychiatric disorders) | 1 | 1 | 6 | NA | NA | NA
Depression suicidal (Psychiatric disorders) | 0 | 0 | 4 | NA | NA | NA
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Major depression (Psychiatric disorders) | 1 | 1 | 7 | NA | NA | NA
Mania (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Mental status changes (Psychiatric disorders) | 0 | 1 | 4 | NA | NA | NA
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 | 0 | 3 | NA | NA | NA
Panic attack (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 2 | NA | NA | NA
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Schizophrenia (Psychiatric disorders) | 0 | 0 | 2 | NA | NA | NA
Somatic symptom disorder (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Substance abuse (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Substance dependence (Psychiatric disorders) | 0 | 1 | 1 | NA | NA | NA
Substance use disorder (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 3 | NA | NA | NA
Suicidal ideation (Psychiatric disorders) | 2 | 4 | 9 | NA | NA | NA
Suicide attempt (Psychiatric disorders) | 1 | 4 | 9 | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 16 | NA | NA | NA
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 0 | 1 | NA | NA | NA
Bladder trabeculation (Renal and urinary disorders) | 1 | 0 | 1 | NA | NA | NA
Calculus urethral (Renal and urinary disorders) | 0 | 0 | 1 | NA | NA | NA
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 2 | NA | NA | NA
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 4 | NA | NA | NA
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 1 | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 1 | 3 | NA | NA | NA
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 3 | NA | NA | NA
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 1 | NA | NA | NA
Nephritic syndrome (Renal and urinary disorders) | 0 | 0 | 1 | NA | NA | NA
Nephrolithiasis (Renal and urinary disorders) | 3 | 2 | 31 | NA | NA | NA
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1 | NA | NA | NA
Renal colic (Renal and urinary disorders) | 0 | 1 | 3 | NA | NA | NA
Renal cyst (Renal and urinary disorders) | 0 | 0 | 2 | NA | NA | NA
Renal failure (Renal and urinary disorders) | 0 | 1 | 3 | NA | NA | NA
Renal haematoma (Renal and urinary disorders) | 0 | 1 | 1 | NA | NA | NA
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | NA | NA | NA
Renal injury (Renal and urinary disorders) | 1 | 0 | 2 | NA | NA | NA
Renal mass (Renal and urinary disorders) | 1 | 0 | 3 | NA | NA | NA
Ureterolithiasis (Renal and urinary disorders) | 2 | 1 | 14 | NA | NA | NA
Urethral obstruction (Renal and urinary disorders) | 0 | 0 | 1 | NA | NA | NA
Urinary bladder rupture (Renal and urinary disorders) | 0 | 0 | 1 | NA | NA | NA
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 0 | 0 | 3 | NA | NA | NA
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 2 | NA | NA | NA
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 2 | NA | NA | NA
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 21 | NA | NA | NA
Breast disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Breast hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 1 | NA | NA | NA
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 4 | NA | NA | NA
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 4 | NA | NA | NA
Feminisation acquired (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | 2 | NA | NA | NA
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 3 | NA | NA | NA
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 | 0 | 1 | NA | NA | NA
Ovarian mass (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 2 | NA | NA | NA
Premature menopause (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Prostatic disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 3 | NA | NA | NA
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 2 | NA | NA | NA
Testicular torsion (Reproductive system and breast disorders) | 0 | 1 | 1 | NA | NA | NA
Uterine disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1 | NA | NA | NA
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | NA | NA | NA
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | NA | NA | NA
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 18 | NA | NA | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 9 | NA | NA | NA
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 25 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 9 | NA | NA | NA
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | NA | NA | NA
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | NA | NA | NA
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | NA | NA | NA
Pleural mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | NA | NA | NA
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 50 | NA | NA | NA
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | NA | NA | NA
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | NA | NA | NA
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | NA | NA | NA
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | NA | NA | NA
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | NA | NA | NA
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 7 | NA | NA | NA
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Tonsillar ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | NA | NA | NA
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | NA | NA | NA
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | NA | NA | NA
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | NA | NA | NA
Miscarriage of partner (Social circumstances) | 0 | 0 | 3 | NA | NA | NA
Organ donor (Social circumstances) | 0 | 0 | 2 | NA | NA | NA
Physical assault (Social circumstances) | 0 | 1 | 2 | NA | NA | NA
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 4 | NA | NA | NA
Aortic aneurysm (Vascular disorders) | 0 | 0 | 2 | NA | NA | NA
Aortic stenosis (Vascular disorders) | 1 | 0 | 5 | NA | NA | NA
Arteriosclerosis (Vascular disorders) | 0 | 0 | 5 | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 4 | 2 | 38 | NA | NA | NA
Embolism venous (Vascular disorders) | 1 | 0 | 1 | NA | NA | NA
Haematoma (Vascular disorders) | 1 | 0 | 1 | NA | NA | NA
Hypertension (Vascular disorders) | 2 | 2 | 6 | NA | NA | NA
Hypertensive crisis (Vascular disorders) | 1 | 0 | 3 | NA | NA | NA
Hypertensive emergency (Vascular disorders) | 0 | 0 | 3 | NA | NA | NA
Hypertensive urgency (Vascular disorders) | 1 | 0 | 3 | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 1 | 5 | NA | NA | NA
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | NA | NA | NA
Leriche syndrome (Vascular disorders) | 0 | 0 | 1 | NA | NA | NA
Lymphoedema (Vascular disorders) | 0 | 0 | 2 | NA | NA | NA
May-Thurner syndrome (Vascular disorders) | 0 | 0 | 1 | NA | NA | NA
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 3 | NA | NA | NA
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 3 | NA | NA | NA
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 1 | NA | NA | NA
Peripheral artery aneurysm rupture (Vascular disorders) | 0 | 0 | 1 | NA | NA | NA
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1 | NA | NA | NA
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 2 | NA | NA | NA
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 2 | NA | NA | NA
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | NA | NA | NA
Peripheral venous disease (Vascular disorders) | 0 | 0 | 1 | NA | NA | NA
Phlebitis (Vascular disorders) | 0 | 0 | 1 | NA | NA | NA
Shock (Vascular disorders) | 0 | 0 | 2 | NA | NA | NA
Thrombophlebitis (Vascular disorders) | 0 | 0 | 2 | NA | NA | NA
Thrombosis (Vascular disorders) | 0 | 0 | 1 | NA | NA | NA
Varicose vein (Vascular disorders) | 0 | 1 | 3 | NA | NA | NA
Vasospasm (Vascular disorders) | 0 | 0 | 1 | NA | NA | NA
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 1 | NA | NA | NA
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 3 | NA | NA | NA
Pancreatolithiasis (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Smear cervix abnormal (Investigations) | 0 | 1 | 0 | NA | NA | NA
Brain stem stroke (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Aggression (Psychiatric disorders) | 1 | 0 | 0 | NA | NA | NA
Thrombophlebitis of the right upper limb cephalic vein (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase: Ad26.COV2.S 5*10^10 vp (N=3356) | Double-blind Phase: Placebo (N=3380) | Combined Double-blind and Open-label Phase: All Participants (N=0) | OL Phase: Ad26.COV2.S 5*10^10 vp + Ad26.COV2.S 5*10^10 vp Booster (N=22213) | Open Label Phase: mRNA 2 Dose Schedule + Ad26.COV2.S 5*10^10 vp Booster (N=613) | OL Phase: Non-mRNA Any Schedule +Ad26.COV2.S vp Booster OR mRNA Other Schedule +Ad26.COV2.S Booster (N=943)
Nausea(Solicited) (Gastrointestinal disorders) | 550 | 363 | NA | 968 | 35 | 67
Chills (General disorders) | 70 | 22 | NA | 20 | 3 | 3
Fatigue(Solicited) (General disorders) | 1420 | 829 | NA | 2589 | 115 | 155
Pyrexia(Solicited) (General disorders) | 250 | 12 | NA | 169 | 20 | 16
Vaccination site erythema (Solicited) (General disorders) | 246 | 134 | NA | 325 | 12 | 27
Vaccination site pain(Solicited) (General disorders) | 1781 | 595 | NA | 3702 | 134 | 201
Vaccination site swelling(Solicited) (General disorders) | 198 | 51 | NA | 316 | 11 | 21
Myalgia(Solicited) (Musculoskeletal and connective tissue disorders) | 1246 | 494 | NA | 2140 | 105 | 126
Headache (Solicited) (Nervous system disorders) | 1454 | 900 | NA | 2220 | 97 | 130
Fatigue (General disorders) | 48 | 70 | NA | 153 | 5 | 21
Headache (Nervous system disorders) | 63 | 70 | NA | 182 | 4 | 17

LIMITATIONS AND CAVEATS:
Safety results are reported in AE section, hence not repeated again in OM section. As pre-specified in statistical analysis plan, data of efficacy OMs for OL booster phase was not collected and analyzed. As clinical development program has moved from "Development" to "Life cycle management" phase, scope and extent of open label analysis was reduced. Hence, data was not collected and analyzed for OMs of platelet count, Biomarkers With SARS-CoV-2 Infection & COVID-19 Severity Using RNA Sequencing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (3):
  • Study Protocol (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT04505722/Prot_002.pdf
  • Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT04505722/SAP_003.pdf
  • Informed Consent Form (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT04505722/ICF_004.pdf